CLINICAL TRIAL: NCT05966675
Title: Physiologic Cardiac Pacing to Prevent Left Ventricular Dysfunction Post Transcatheter Aortic Valve Implantation
Brief Title: Physiologic Cardiac Pacing to Prevent Left Ventricular Dysfunction Post TAVI
Acronym: PACE-4-TAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022/ABM/03/00049
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Atrioventricular Block, Second and Third Degree
Keywords: Pacemaker; Transcatheter Aortic Valve Replacement; Conduction System Pacing (CSP); Atrioventricular Block; Congestive Heart Failure; Bradycardia
MeSH Terms: conditions — Atrioventricular Block; Neoplasm Metastasis; Heart Failure; Bradycardia | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to the intervention and control groups. In the control group, the type of ventricular pacing will depend on the left ventricular ejection fraction (LVEF): 1) RVP is planned in the group of patients with LVEF ≥40%, 2) BVP is planned in the group of patients with LVEF <40%, following current ESC guidelines.
Who Masked: Participant
Masking Description: Patient will be blind to type of intervention. Due to a need of method-specific use of hardware and tailored programming of cardiac devices, medical staff is impossible to blind. The inability to blind affects also echocardiographists and anyone performing device interrogation as significant differences in number and localisation of pacing leads, their electrical parameters and pacemaker settings are inherently different in studied arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conduction System Pacing (Experimental): Patients who receive Conduction System Pacing in form of Left Bundle Branch Area Pacing or His Bundle Pacing.
  Interventions: Device: conduction system pacing
- Standard Pacing Method (Active Comparator): Patients who receive currently standard pacing method with exact type of ventricular pacing depending upon left ventricular ejection fraction (LVEF): right ventricular pacing in case of LVEF >= 40% or biventricular pacing if LVEF is determined to be less than 40%, as per current ESC guidelines.
  Interventions: Device: right ventricular or biventricular pacing

INTERVENTIONS:
Device: conduction system pacing — Implantation of cardiac implantable electronic device (CIED) with conduction system pacing (left bundle branch area pacing or his bundle pacing).
  Arms: Conduction System Pacing
Device: right ventricular or biventricular pacing — Implantation of cardiac implantable electronic device with right ventricular or biventricular pacing according to left ventricular ejection fraction and current ESC guidelines.
  Arms: Standard Pacing Method

SUMMARY:
The study aims to compare permanent Conduction System Pacing (CSP) with the standard therapy - Right Ventricular Pacing (RVP) or Biventricular Pacing (BVP) - in preventing the development and progression of symptomatic Chronic Heart Failure (CHF) and improving survival in patients after Transcatheter Aortic Valve Implantation (TAVI).

DETAILED DESCRIPTION:
A multicenter randomized controlled head-to-head trial was planned to compare the effects of permanent pacemaker implantation (PPMI) using CSP (study intervention) with currently standard therapy - RVP or BVP (control group). The study population will consist of patients hospitalized after TAVI complicated with high-degree persistent atrioventricular (AV) block or newly developed complex AV or intraventricular conduction disturbances, qualified for PPMI within 30 days after surgery, following the 2021 European Society of Cardiology (ESC) guidelines on cardiac pacing and cardiac resynchronization therapy.

ELIGIBILITY:
Inclusion Criteria:

1. transcatheter aortic valve implantation (TAVI) in up to 30 days before qualification to pacemaker implantation
2. Fulfilled criteria for permanent pacemaker implantation according do 2021 ESC guidelines
3. Written informed consent
4. Age of at least 18 years

Exclusion Criteria:

1. Permanent pacemaker implantation before TAVI procedure
2. The occurrence of conduction disturbances more than 30 days after TAVI procedure
3. No written informed consent
4. Inability to obtain informed consent from participant
5. Predicted inability to obtain cooperation from patient during observation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Heart Failure Hospitalization | 12 months
  Hospitalization due to heart failure as a main reason
All-cause death | 12 months
  Death from any cause

SECONDARY OUTCOMES:
Change in exercise capacity | 24 months
  Improvement or deterioration in exercise capacity assessed as a change of ≥1 New York Heart Association (NYHA) functional class or a change in 6-Minute Walk Test (6MWT) distance by 55m or more
Response to Cardiac Resynchronization Therapy (CRT) | 24 months
  Meeting the echocardiographic criteria of response to CRT defined as a decrease in Left Ventricular End Systolic Volume by ≥15% or an increase in Left Ventricular Ejection Fraction by ≥5% from the baseline values
Pacing-Induced Cardiomyopathy (PICM) | 24 months
  Pacing-related CHF meeting the echocardiographic criteria of PICM defined as a decrease in LVEF by >=10% to the absolute value of <50%
Change in global longitudinal strain (GLS) | 24 months
  An increase in GLS value of 20 absolute percentage points from baseline or an increase above -16%.
Atrial Fibrillation (AF) episodes | 24 months
  Occurrence of the first episode of AF in a patient with no previous history of atrial fibrillation (AF).
Atrial High Rate Episodes (AHRE) in pacemaker recordings | 24 months
  Occurrence or change of the burden of AHRE events in the records from the CIED.
Change in the concentration of the N-terminal pro-brain natriuretic peptide (NT-proBNP) | 24 months
  pl/mL
Change in Quality of Life | 24 months
  Assessed with Short Form Health Survey (SF-36): 0 to 100; low QoL to high QoL - better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof S. Gołba, MD PhD, Study Chair — Silesian Medical University in Katowice
Locations (1):
- Medical University of Silesia in Katowice, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Background] Shimony A, Eisenberg MJ, Filion KB, Amit G. Beneficial effects of right ventricular non-apical vs. apical pacing: a systematic review and meta-analysis of randomized-controlled trials. Europace. 2012 Jan;14(1):81-91. doi: 10.1093/europace/eur240. Epub 2011 Jul 27. PMID 21798880
- [Background] Daubert JC, Ritter P, Le Breton H, Gras D, Leclercq C, Lazarus A, Mugica J, Mabo P, Cazeau S. Permanent left ventricular pacing with transvenous leads inserted into the coronary veins. Pacing Clin Electrophysiol. 1998 Jan;21(1 Pt 2):239-45. doi: 10.1111/j.1540-8159.1998.tb01096.x. PMID 9474680
- [Background] Dandamudi G, Vijayaraman P. How to perform permanent His bundle pacing in routine clinical practice. Heart Rhythm. 2016 Jun;13(6):1362-6. doi: 10.1016/j.hrthm.2016.03.040. Epub 2016 Mar 22. No abstract available. PMID 27016475
- [Background] Huang W, Chen X, Su L, Wu S, Xia X, Vijayaraman P. A beginner's guide to permanent left bundle branch pacing. Heart Rhythm. 2019 Dec;16(12):1791-1796. doi: 10.1016/j.hrthm.2019.06.016. Epub 2019 Jun 22. No abstract available. PMID 31233818
- [Background] Jastrzebski M, Moskal P, Bednarek A, Kielbasa G, Vijayaraman P, Czarnecka D. Programmed His Bundle Pacing: A Novel Maneuver for the Diagnosis of His Bundle Capture. Circ Arrhythm Electrophysiol. 2019 Feb;12(2):e007052. doi: 10.1161/CIRCEP.118.007052. PMID 30707037
- [Background] Jastrzebski M, Moskal P, Bednarek A, Kielbasa G, Kusiak A, Sondej T, Bednarski A, Vijayaraman P, Czarnecka D. Programmed deep septal stimulation: A novel maneuver for the diagnosis of left bundle branch capture during permanent pacing. J Cardiovasc Electrophysiol. 2020 Feb;31(2):485-493. doi: 10.1111/jce.14352. Epub 2020 Jan 20. PMID 31930753
- [Background] Nazif TM, Dizon JM, Hahn RT, Xu K, Babaliaros V, Douglas PS, El-Chami MF, Herrmann HC, Mack M, Makkar RR, Miller DC, Pichard A, Tuzcu EM, Szeto WY, Webb JG, Moses JW, Smith CR, Williams MR, Leon MB, Kodali SK; PARTNER Publications Office. Predictors and clinical outcomes of permanent pacemaker implantation after transcatheter aortic valve replacement: the PARTNER (Placement of AoRtic TraNscathetER Valves) trial and registry. JACC Cardiovasc Interv. 2015 Jan;8(1 Pt A):60-9. doi: 10.1016/j.jcin.2014.07.022. PMID 25616819
- [Background] Xi Z, Liu T, Liang J, Zhou YJ, Liu W. Impact of postprocedural permanent pacemaker implantation on clinical outcomes after transcatheter aortic valve replacement: a systematic review and meta-analysis. J Thorac Dis. 2019 Dec;11(12):5130-5139. doi: 10.21037/jtd.2019.12.02. PMID 32030230
- [Background] Xu S, Zhang E, Qian Z, Sun J, Zou F, Wang Y, Hou X, Zou J. Mid- to Long-Term Clinical and Echocardiographic Effects of Post-procedural Permanent Pacemaker Implantation After Transcatheter Aortic Valve Replacement: A Systematic Review and Meta-Analysis. Front Cardiovasc Med. 2022 Jun 28;9:911234. doi: 10.3389/fcvm.2022.911234. eCollection 2022. PMID 35837611
- [Background] Fadahunsi OO, Olowoyeye A, Ukaigwe A, Li Z, Vora AN, Vemulapalli S, Elgin E, Donato A. Incidence, Predictors, and Outcomes of Permanent Pacemaker Implantation Following Transcatheter Aortic Valve Replacement: Analysis From the U.S. Society of Thoracic Surgeons/American College of Cardiology TVT Registry. JACC Cardiovasc Interv. 2016 Nov 14;9(21):2189-2199. doi: 10.1016/j.jcin.2016.07.026. PMID 27832844